CLINICAL TRIAL: NCT00994799
Title: Comparison of the Effect of Intravitreal Ranibizumab Injections Compared to Macular Grid-pattern Laser Therapy for the Symptomatic Treatment of Diabetic Macular Edema (a Randomized, Controlled, Phase III Trial)
Brief Title: Comparison of Intravitreal Ranibizumab and Macular Grid-pattern Laser for Treatment of Diabetic Macular Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Collaborators: Semmelweis University (Other); Csolnoky Ferenc County Hospital (Unknown)
Responsible Party: Lajos Kolozsvari Dr Prof, University of Szeged Department of Ophthalmology
Other Study IDs: CRFB002AHU04T; CRFB002DHU06T
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ranibizumab group: patients receiving intravitreal ranibizumab for diabetic macular edema
  Interventions: Drug: ranibizumab
- laser: patients receiving macular grid-pattern laser therapy
  Interventions: Radiation: macular grid-pattern laser

INTERVENTIONS:
Drug: ranibizumab — 10mg/ml intravitreal injection
  Other Names: Lucentis
  Groups: ranibizumab group
Radiation: macular grid-pattern laser — macular grid-pattern laser therapy
  Other Names: macular laser
  Groups: laser

SUMMARY:
This study investigates the hypothesis that ranibizumab injection given into the eye is an efficacious and safe treatment option applied for swelling of the macula (site of sharp vision) in diabetes.

DETAILED DESCRIPTION:
This is a randomized, controlled, three-center trial to assess the efficacy and safety of intravitreal ranibizumab injections in diabetic macular edema. Comparator arm consists of patients receiving macular grid-pattern laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female type I or II diabetic patients over 18 years of age
* Diagnosis of DME secondary to diabetic retinopathy and decrease in vision is due to DME and not due to other causes in the opinion of the investigator
* Patients who have a BCVA score between 78 and 39 letters in the study eye using ETDRS-like visual acuity charts at a testing distance of 4 meters
* Expectation by the investigator that patient will potentially benefit from laser treatment or ranibizumab treatment
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Active intraocular inflammation, any active infection or history of uveitis
* Uncontrolled glaucoma or neovascularization of the iris in the study eye
* Structural damage within 0.5 disc diameter of the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), epiretinal membrane involving fovea or organized hard exudate plaques
* Concurrent disease in the study eye that could compromise visual acuity or prevent the improvement of visual acuity (including diabetic proliferative retinopathy) or require medical or surgical intervention during the study period, including cataract, retinal vascular occlusion, retinal detachment, macular hole or choroidal neovascularization of any cause
* Panretinal laser photocoagulation in the study eye within 6 months prior to or during the study or focal/grid laser photocoagulation in the study eye within 3 months prior to study entry
* Treatment with anti-angiogenic drugs (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc) or intravitreal corticosteroids in the study eye within 3 months prior to randomization
* Any intraocular surgery in the study eye within 3 months prior to randomization
* History of vitrectomy in the study eye
* Ocular conditions in the study eye that require chronic concomitant therapy with topical ocular or systemically administered corticosteroids
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes patients having clinically significant macular edema due to diabetic retinopathy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Mean change in best corrected visual acuity | 12 months

SECONDARY OUTCOMES:
Mean change in retinal thickness as assessed with OCT | 12 months
Change in the extension of foveal avascular zone, foveal thickness and macular volume by FA and OCT, respectively. | 12 months
Change in retinal function (color vision,contrast sensitivity, multifocal ERG) | 12 months
Rate of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Kolozsvari, prof, Principal Investigator — Szeged University
Locations (3):
- Hungary (3):
  - Semmelweis University Department of Ophthalmology, Budapest
  - University of Szeged, Medical and Pharmaceutical Center, Department of Ophthalmology, Szeged
  - Csolnoky Ferenc County Hospital Dept of Ophthalmolgy, Veszprém